CLINICAL TRIAL: NCT05763979
Title: Assesment of the Change in Consumer Behaviours to Afford the Dietary Cost According to Food Security Status and Choice Motives
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Mehmet HAYDAROGLU, Research Assistant, Hacettepe University
Other Study IDs: TIF-Con
Record Dates: First submitted 2023-03-01; First posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Food Selection; Consumer Behavior; Healthy Nutrition
Keywords: Food security; Food choice motives; Food inflation; Healthy Diet's Cost
MeSH Terms: conditions — Food Preferences; Consumer Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to assement of the change in consumer behaviours during the food inflation period in order to afford the dietary cost according to food security status and food choice motives. The study was planned in four stages. 1) First stage is adapting the Single-item Food Choice Questionnaire to Turkish society and to make its validity and reliability in Turkish. 2) The Impact of Food Inflation on Consumer Behavioural Change (TIF-Con) scale will be developed. 3) Observational cross-sectional data collection including these surveys will be carried out. 4) The Cost of the Recommended Diet (CoRD) will be calculated by collecting data simultaneously with the fieldwork. Hypotheses will be tested in line with the findings obtained.

DETAILED DESCRIPTION:
The reliability and validity of the Single-item Food Choice Questionnaire was planned in eight stages. 1) Translation into Target Language 2) Synthesis of translations 3) Back translation to Original Language 4) Expert assessment 5) Pilot study 6) Reporting 7) Testing 8) Retesting. The development of the Impact of Food Inflation on Consumer Behavioural Change (TIF-Con) scale was planned in eight stages too. 1) Generating an item pool 2) Determining the format for measurement 3) Initial item pool reviewed by experts 4) Pretesting 5) Optimizing scale length 6) Testing 7) Retesting 8) Reporting. A cross-sectional survey will be conducted by questioning food security and socioeconomic status, along with the developed TIF-Con and the adapted food choice questionnaire. This stage will be combined with the sixth stage of scale development in order to act economically. Simultaneously, the CoRD will be calculated with the collection of food prices with fieldwork and the recommendations of the offical Turkey's dietary guideline. The obtained results will be analyzing to assesment of the change in consumer behaviours during the food inflation period in order to afford the dietary cost according to food security status and food choice motives.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-65
* Who volunteered to participate in the study
* Adult individuals who have access to the Internet and agreed to participate in the study
* Native language being Turkish
* Living in Turkey at least five years

Exclusion Criteria:

* Those with a disease that requires a specific diet
* Inability to use a computer, tablet or mobile phone
* Native language not being Turkish
* Those who have not lived in Turkey for at least five years

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People who live in Turkey and meeting the inclusion criteria and volunteered to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Food choice motives | 03.15.2023
  The identifying of consumers' food choice motives with using the Single-item Food Choice Questionnaire
The Impact of Food Inflation on Consumer Behavioural Change | 04.15.2023
  The identifying of the change in consumer behaviours during the food inflation period

SECONDARY OUTCOMES:
Consumer Behavioural Changes' Differences | 06.15.2023
  Consumer behavioural changes' differences in afford the dietary cost according to food security status and food choice motives

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Nutrition and Dietetics Department, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided